CLINICAL TRIAL: NCT07140536
Title: Einfluss Von Laufbändern für Büroarbeitsplätze Auf Ergonomie, Heizenergiebedarf, Leistungsfähigkeit Sowie Rücken- Und Kardiometabolische Gesundheit
Brief Title: The Impact of Treadmills and Cooler Environments for Office Workplaces on Ergonomics, Heating Energy Requirements, Performance, as Well as Back and Cardiometabolic Health
Acronym: ELBEngLück
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Jan-Frieder Harmsen, Principal Investigator, RWTH Aachen University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EK 25-134
Record Dates: First submitted 2025-08-11; First posted 2025-08-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy Male and Female Subjects
Keywords: sit less; break sitting time; ergonomics; cardiometabolic health; thermal comfort; office treadmill; glucose control; blood pressure; attention
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sedentary activity at standard room temperature (23°C) (Experimental): Sedentary activity at standard room temperature (23°C)
  Interventions: Other: Environmental temperature; Behavioral: Physical activity
- Walking activity at standard room temperature (23°C) (Experimental): Walking activity at standard room temperature (23°C)
  Interventions: Other: Environmental temperature; Behavioral: Physical activity
- Sedentary activity at lowered room temperature (19°C) (Experimental): Sedentary activity at lowered room temperature (19°C)
  Interventions: Other: Environmental temperature; Behavioral: Physical activity
- Walking activity at lowered room temperature (19°C) (Experimental): Walking activity at lowered room temperature (19°C)
  Interventions: Other: Environmental temperature; Behavioral: Physical activity

INTERVENTIONS:
Other: Environmental temperature — The office is day is spent in 19 or 23°C room temperature from 08:30AM to 04:30PM.
Behavioral: Physical activity — From 08:30AM to 04:30PM, the office is day is spent either fully sedentary or interspersed with light walking on a treadmill (60 min at 10:00AM, 15 min at 01:00PM, 15 min at 02:00PM, 15 min at 03:00PM, 15 min at 04:00PM).

SUMMARY:
The aim of the project is to gain insights into the effects of treadmills at a standing desk and reduced room temperature on back and cardiometabolic health, cognitive performance, thermal comfort, and the associated heating energy requirements of buildings.

Healthy young men and women will spend four consecutive days in a controlled laboratory office environment after a baseline visit. During the baseline visit, volunteers are familiarized with the treadmill and start wearing a continuous glucose monitor. The four consecutive laboratory office days are each scheduled from 8:30AM to 04:30PM. In a randomized order, participants the first two office days either at 19°C or 23°C room temperature. The first office day of each temperature conditions is spent only sedentary, while for the second one is regularly interrupted with light walking on the treadmill. Otherwise, the daily routine and test battery will be exactly the same between days, including a standardized breakfast and lunch meal, an attention task in the morning, and frequent subjective thermal comfort ratings and blood pressure measurements. Interstitial glucose as well as heart rate and heart rate variability will be continuously monitored through wearable devices. Treadmill walking will be videorecorded.

DETAILED DESCRIPTION:
This is a controlled intervention study with a crossover design. Participants are assigned to different conditions in which they perform both sedentary and walking desk activities at different room temperatures.

Intervention conditions:

I: Sedentary activity at standard room temperature (23°C) II: Walking activity at standard room temperature (23°C) III: Sedentary activity at lowered room temperature (19°C) IV: Walking activity at lowered room temperature (19°C)

Each condition is carried out over a defined period, with corresponding 24-hour washout periods between conditions to minimize carry-over effects.

Participants are expected to attend a total of five in-person appointments at the indoor climate laboratory of the Chair of Building Services Engineering at RWTH Aachen University. On Day 0, an introduction to the local conditions will take place before the actual study week begins, and the continuous glucose monitor is individually placed on the upper arm. In the following study week, four consecutive experimental study days are planned. Participants will go through two different scenarios: Six participants will first experience a warm exposure for two days, followed by a cold exposure for two days, while the other six will start with a cold exposure and end with the warm exposure. Allocation of participants to the two sequences of the four experimental conditions (Sequence 1: I-II-III-IV; Sequence 2: III-IV-I-II) is performed using stratified block randomization. A computer-generated randomization procedure is used to ensure that participants are evenly distributed between both sequences. Randomization is carried out before the first test session. To ensure a balanced gender distribution, ideally three men and three women will start with Sequence 1, and three men and three women with Sequence 2.

Participants meet at 8:30 a.m. at the indoor climate laboratory of the Chair of Building Services Engineering and begin preparations, during which the required sensors for data collection are attached. The clothing level of participants will be approximately 0.8 clo for all conditions (DIN EN ISO 9920, 2009-10: Ergonomics of the thermal environment - Estimation of the thermal insulation and evaporative resistance of a clothing ensemble). In practice, this results in the following clothing requirement, which will be communicated to participants on Day 0: underwear, socks, shoes, long trousers, T-shirt/undershirt, and a long-sleeved shirt.

Each of the four laboratory office days follows in principle the same time course. From 08:30AM onwards, a chest-worn heart rate monitor belt is started to be worn. At 9:00AM, a breakfast meal (standardized liquid meal) will be taken under controlled conditions. This is followed at 10:00AM by the first activity phase: participants in the walking conditions walk for one hour on the treadmill, while those in the sedentary conditions perform seated work and remain seated throughout. From 10 to 11:00AM, participants will perform an attention task on a computer. At 11:00AM, a recovery phase begins, during which participants complete a standardized questionnaires for subjective ratings. At 12:30, lunch is served (e.g., bread, fruit, and cereal bars). Starting at 1:00PM, four consecutive short activity periods take place every hour: for 15 minutes each, participants in the walking conditions walk on the treadmill, while those in the sedentary conditions continue to sit, interspersed with 45 min sitting for all conditions. At 4:15PM after the last walking activity, a final survey is conducted, during which a concluding questionnaire is completed to evaluate the overall experience and any changes in well-being. At regular intervals over each laboratory office day, participants will be asked to rate their thermal comfort on digital scales and blood pressure will be measured preceding and following walking periods. Each laboratory day officially ends at 4:30PM with the removal of sensors and the participants' departure. Only the continuous glucose monitor will only be removed on the fourth and last test day.

ELIGIBILITY:
Inclusion Criteria:

* Physically active, healthy test subjects
* Participants who are able to understand the research project
* Adult test volunteers (aged >18 and <40)
* German language skills at B2-C2 level

Exclusion Criteria:

* An implanted pacemaker
* Participants who are unable to give consent/participants with a legal representative
* Age under 18 or over 40
* Pregnant participants
* Participants with a BMI >28
* Participants with underlying diseases with significant functional limitations (e.g., rheumatoid arthritis, diabetes mellitus, high blood pressure)
* Reading and/or spelling disorders or combined disorders of scholastic skills (ICD-10 F81.0 - F81.3)
* Participants with a possible SARS-CoV-2 infection will be excluded from the study for the duration of the infection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Subjective thermal comfort rating | At regular intervals over each of the four laboratory office days
Interstitial glucose levels | Continuously sampled every 15 min over all four laboratory office days
  Interstitial glucose levels measured by continuous glucose monitors
Working memory assessed by the TAP (Zimmermann & Fimm, 2002) n-back task | 10:00-11:00 AM during each of the four laboratory office days
  Participants view sequences of numbers and indicate whether the current number matches one presented one or two steps earlier. Outcome variables are accuracy (% correct) and reaction time (ms).
Divided attention assessed by the TAP (Zimmermann & Fimm, 2002) divided attention task | 10:00-11:00 AM during each of the four laboratory office days
  Participants simultaneously perform a visual and an auditory discrimination task. Outcome variables are reaction time (ms) and error rates.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | at 09:00, 11:00, 12:30, 14:30 and 16:00 over all four laboratory office days
  Manually measured via automated blood pressure cuffs
Heart rate | continuously from 08:30AM to 04:30PM over all four laboratory office days
  assessed continuously via chest-worn belts
Heart rate variability | continuously from 08:30AM to 04:30PM over all four laboratory office days
  assessed continuously via chest-worn belts
Skin temperature | continuously from 08:30AM to 04:30PM over all four laboratory office days
  via adhesive thermal sensors placed on different skin regions
Cognitive flexibility assessed by the TAP (Zimmermann & Fimm, 2002) task-switching module | 10:00-11:00 AM during each of the four laboratory office days
  Participants alternate their responses to different types of visual stimuli based on changing task rules. Outcome variables are reaction time (ms) and number of errors.
Intrinsic and phasic alertness assessed by the TAP (Zimmermann & Fimm, 2002) alertness task | 10:00-11:00 AM during each of the four laboratory office days
  Participants respond to visual stimuli on a screen with and without an auditory warning cue. Outcome variables are reaction time (ms) and error rates.
Sustained attention assessed by the TAP (Zimmermann & Fimm, 2002) sustained attention task | 10:00-11:00 AM during each of the four laboratory office days
  Participants monitor a continuous stream of visual stimuli and respond when the current item matches the previous one in certain features. Outcome variables are reaction time (ms), omission errors, and commission errors.
Hip joint angles and dynamics during gait assessed by sagittal plane video analysis | During the walking period between 10:00-11:00 AM on each of the 4 laboratory days
  Range of motion, angular displacement, and angular velocity of the hip joint will be extracted from sagittal plane video recordings during walking.
Knee joint angles and dynamics during gait assessed by sagittal plane video analysis | During the walking period between 10:00-11:00 AM on each of the 4 laboratory days
  Range of motion, angular displacement, and angular velocity of the knee joint will be extracted from sagittal plane video recordings during walking.
Spinal joint angles and dynamics during gait assessed by sagittal plane video analysis | During the walking period between 10:00-11:00 AM on each of the 4 laboratory days
  Range of motion, angular displacement, and angular velocity of the spine will be extracted from sagittal plane video recordings during walking.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Frieder Harmsen, PhD, Principal Investigator — RWTH Aachen University
Locations (1):
- University hospital at RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The study protocol can be requested via email to study officials.
Supporting Information: Study Protocol
Time Frame: The study protocol is available from the 11th of August 2025 onwards for at least 5 years.
Access Criteria: The study protocol can be requested via email to study officials.